CLINICAL TRIAL: NCT06152809
Title: A Phase 1 Study of Cytokine-induced Memory-like (CIML) NK Cells With Venetoclax as Consolidation Therapy in AML
Brief Title: CIML NK Cells With Venetoclax for AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Evan Chen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-534
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Recurrent; Leukemia; Leukemia, Myeloid
Keywords: Acute Myeloid Leukemia; Acute Myeloid Leukemia Recurrent; Leukemia; Leukemia, Myeloid
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Leukemia, Myeloid | interventions — Interleukin-2; aldesleukin; venetoclax

STUDY DESIGN:
Intervention Model Description: One group of patients, two dose levels (arms)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Dose Level 0 (Experimental): A maximum tolerated dose (MTD) will be established, and dosage will start at dose level 0. 5-10 participants at dose level 0 will complete:
  * Baseline visit.
  * Bone marrow biopsies: at screening visit #2, end of treatment, and at discretion of PI.
  * Days -6 through -2: predetermined doses of standard-of-care lymphodepleting chemotherapy.
  * Day 0: Predetermined dose of CIML NK cells 1x daily. Hospitalization for up to 3 to 4 weeks for CIML NK infusion.
  * Days 0 through 12: Predetermined dose of IL-2 1x daily every other day for up to 5 doses.
  * Day 7 through Day 21: Predetermined dose of Venetoclax 1 x daily.
  * If ≤1 dose-limiting toxicities (DLTs) are observed, this dose will be the MTD, and 5 additional participants will be enrolled.
  * Follow-up visits: Days 42, 60, 100 and months 6, 9, and 12.
  Interventions: Biological: Cytokine-Induced Memory-like Natural Killer Cells; Biological: Interleukin-2; Drug: Venetoclax
- Cohort 1: Dose Level -1 (Experimental): De-escalation to dose level -1 will be conducted per protocol if DLTs occur in Cohort 1 dose Level 0. Participants will complete:
  * Baseline visit.
  * Bone marrow biopsies: at screening visit #2, end of treatment, and at discretion of PI.
  * Days -6 through -2: predetermined doses of standard-of-care lymphodepleting chemotherapy.
  * Day 0: Predetermined dose of CIML NK cells 1x daily. Hospitalization for up to 3 to 4 weeks for CIML NK infusion.
  * Days 0 through 12: Predetermined dose of IL-2 1x daily every other day for up to 5 doses.
  * Day 7 through Day 21: Predetermined dose of Venetoclax 1 x daily.
  * Follow-up visits: Days 42, 60, 100 and months 6, 9, and 12.
  Interventions: Biological: Cytokine-Induced Memory-like Natural Killer Cells; Biological: Interleukin-2; Drug: Venetoclax

INTERVENTIONS:
Biological: Cytokine-Induced Memory-like Natural Killer Cells — Allogeneic, cytokine induced memory-like natural killer cells, via intravenous infusion per protocol.
  Other Names: CIML NK Cells
Biological: Interleukin-2 — Recombinant, human glycoprotein, single-use 22 MIU vials, via subcutaneous (under the skin) injection per protocol.
  Other Names: Aldesleukin, Proleukin, IL-2
Drug: Venetoclax — Selective inhibitor of BCL-2 protein, 10, 50, or 100 mg tablets, via orally per standard-of-care.
  Other Names: C45H50ClN7O7S

SUMMARY:
The purpose of this research study is to test the safety and to explore the effectiveness of infusing cytokine- induced memory-like (CIML) natural killer (NK) cells in combination with Interleukin-2 (IL-2) and standard-of-care venetoclax as a treatment for Acute Myeloid Leukemia (AML).

Names of the study therapies involved in this study are:

* Lymphodepleting therapy with Fludarabine and Cyclophosphamide prior to CIML NK cell infusion
* CIML NK (a cellular therapy)
* IL-2 (a recombinant, human glycoprotein)
* Venetoclax (a selective inhibitor of BCL-2 protein)

DETAILED DESCRIPTION:
This is an open-label, single center phase I trial combining Cytokine-induced memory-like natural killer (CIML NK) cell therapy with low-dose IL-2 and with venetoclax as consolidation therapy in acute myeloid leukemia (AML).

This is the first time that CIML NK cells in combination with venetoclax will be given to humans.

The U.S. Food and Drug Administration (FDA) has not approved CIML NK cells as a treatment for AML.

The U.S. FDA has not approved IL-2 for AML but it has been approved for other uses.

The U.S. FDA has approved venetoclax as a treatment option for AML.

The research study procedures include screening for eligibility, study treatment visits, electrocardiograms (ECGs), bone marrow biopsies, blood tests, and echocardiograms.

Participants will be followed for up to 1 year after the start of therapy.

It is expected that about 10 people will take part in this research study.

This research is funded by the Leukemia and Lymphoma Society.

ELIGIBILITY:
Inclusion Criteria for Trial Enrollment (Screening Visit #1):

* Diagnosis of acute myeloid leukemia (AML)
* Age ≥ 18 years old
* At time of screening patient is being treated with HMA(azacitidine or decitabine) + venetoclax therapy and has received at least 1 cycle of HMA (azacitidine or decitabine) + venetoclax. Patients can have received other lines of therapy prior to HMA + venetoclax therapy including prior chemotherapy and any prior stem cell transplant, provided that the stem cell transplant is > 6 months prior with no ongoing need for immunosuppressive therapy for active graft-versus-host disease.
* Presence of molecular risk factors for relapse with continued HMA + venetoclax therapy as defined by any of the following present at the time of diagnosis or start of HMA + venetoclax therapy (these do not need to be present at the time the screening BM biopsy):

  * 2022 ELN adverse risk karyotype: t(6;9)(p23.3;q34.1)/DEK::NUP214; t(v;11q23.3)/KMT2A-rearranged; t(9;22)(q34.1;q11.2)/BCR::ABL1; t(8;16)(p11.2;p13.3)/KAT6A::CREBBP; inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2)/ GATA2, MECOM(EVI1), t(3q26.2;v)/MECOM(EVI1)-rearranged; -5 or del(5q); -7; Complex karyotype, monosomal karyotype
  * 2022 ELN adverse risk mutations: Any one of the following mutations: Mutated TP53, ASXL1, BCOR, EZH2, RUNX1, SF3B1, SRSF2, STAG2, U2AF1, and/or ZRSR2
  * Additional mutations associated with acquired resistance to venetoclax: Mutated NRAS, KRAS, FLT3 ITD/TKD
* ECOG performance status ≤2 (see Appendix A)
* Participants must meet the following organ function as defined below:

  * Direct bilirubin: ≤1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then < 3 x ULN)
  * AST(SGOT)/ALT(SGPT): ≤3 x institutional ULN
  * creatinine clearance ≥ 45 mL/min; calculated by the Cockcroft Gault formula
  * oxygen saturation ≥ 90% on room air
  * left ventricular ejection fraction ≥ 40%
* Negative pregnancy test for women of childbearing potential only.
* The effects of CIML NK cells and IL-2 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and until 4 months after the last IL-2 dose administration.
* Participants with current symptoms of cardiac disease should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)
* Subjects must be able to swallow pills.
* No laboratory evidence of ongoing hemolysis in opinion of investigator (demonstration of hemolysis should include a haptoglobin level that is below assay).

Exclusion Criteria for Trial Enrollment (Screening visit #1)

* Prior allogeneic stem cell transplant, organ transplant or donor lymphocyte infusion (DLI), CAR-T cell or NK cell therapy
* Persisting Grade > 1 non hematologic toxicity related to prior therapy; however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease disease requiring any steroids >> the equivalent dose of 10 mg of prednisone or other immunosuppressive therapies at the time of this screening visit (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]) and motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis). Patients with Hashimoto's thyroiditis are eligible to go on study.
* Pregnant women are excluded from this study because of the unknown teratogenic risk of CIML NK cells and IL-2 and with the potential for teratogenic or abortifacient effects by Flu/Cy chemotherapy regimen. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CIML NK cells and IL-2, breastfeeding should be discontinued if the mother is treated on this study.
* HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions with anti-retroviral agents used in this study. In addition, these participants are at increased risk of lethal infections when treated with marrow suppressive therapy.
* Individuals with active uncontrolled hepatitis B or C are ineligible as they are at high risk of lethal treatment-related hepatotoxicity after conditioning therapy.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: 1. History of other malignancy and have had complete remission of disease for at least 2 years; 2. Diagnosed and treated within the past 2 years for: nonmetastatic melanoma, surgically resected (not needing systemic chemotherapy) squamous cell carcinoma of skin and nonmetastatic prostate cancer not needing systemic chemotherapy.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to IL-2 or other agents used in study.
* Participants who are receiving any other investigational agents for this condition
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior history of Grade 2 or higher hemolytic anemia (≥ 2g decrease in hemoglobin plus laboratory evidence of hemolysis) from any cause.

Inclusion Criteria to Start Investigational Treatment Plan (Screening visit #2)

* Patient was eligible for protocol per section 3.1.
* Repeat bone marrow biopsy at this time shows a complete remission (CR) or complete remission with incomplete count recovery (CRi) or morphologic leukemia free state (MLFS) (< 5% blasts) but with presence of measurable residual disease (MRD+). MRD can be determined by either flow cytometry, next generation sequencing or PCR. Patients with only persistent DNMTA, TET2 or ASXL1 mutations will not qualify as MRD+ as these DTA mutations without other comutations are associated with clonal hematopoiesis. OR
* Repeat bone marrow biopsy at this time shows 5-19% residual myeloblasts in the bone marrow by either bone marrow aspirate or core biopsy.
* Confirmed haploidentical or fully HLA-matched related donor that is willing and eligible for non-mobilized collection.
* ECOG performance status ≤2 (see Appendix A)
* Participants must meet the following laboratory and organ function as defined below:

  * Direct bilirubin: ≤1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then < 3 x ULN)
  * AST(SGOT)/ALT(SGPT): ≤3 x institutional ULN
  * creatinine clearance ≥ 45 mL/min; calculated by the Cockcroft Gault formula
  * oxygen saturation ≥ 90% on room air
  * left ventricular ejection fraction (LVEF) ≥ 40%
* No significant change in clinical status that would, in the opinion of the investigator, increase the risk of adverse events associated with CIML NK infusion, (e.g., symptomatic congestive heart failure, unstable angina, cardiac arrhythmia)
* Negative pregnancy test for women of childbearing potential only.
* Subjects must be able to swallow pills.

Exclusion Criteria to Start Investigational Treatment Plan (Screening visit #2)

* No live vaccines within the last 6 months.
* No ongoing or active infections.
* Moderate/strong inhibitors of CYP3A except of antifungal medications (such as posaconazole, voriconazole) which the patient is on and the dose of venetoclax has already been adjusted. These are excluded as moderate/strong inhibitors of CYP3A induce higher drug levels of venetoclax which in turns carry the risk of CIML NK cell elimination.
* The presence of donor-specific antibodies (DSAs) with mean fluorescence intensity (MFI) >1000 using a standard assay in subjects who do not receive a desensitization protocol prior to and during stem cell transplant.

Criteria to Receive Lymphodepletion on Day -5

* Adequate organ function within 24 hours of lymphodepletion as defined below:

  * Direct bilirubin: ≤ 1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then < 3 x ULN)
  * AST (SGOT)/ALT (SGPT): ≤ 3 x institutional ULN
* No significant change in clinical status that would, in the opinion of the investigator, increase the risk of adverse events associated with lymphodepletion, (e.g., significant hypoxemia, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia)
* No evidence of active, uncontrolled infection. Patients receiving antibiotics for an infection may be treated if they have clinically responded to antibiotics. These cases should be reviewed with the study PI before proceeding.
* No live vaccines within the last 6 months

Criteria to Receive CIML NK Infusion

* Adequate organ function within 24 hours of NK cell infusion as defined below:

  * Direct bilirubin: ≤1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then < 3 x ULN)
  * AST(SGOT)/ALT(SGPT): ≤3 x institutional ULN
  * Creatinine clearance ≥ 45 mL/min; calculated by the Cockcroft Gault formula
* No Grade ≥3 non-hematologic toxicities of cyclophosphamide and fludarabine conditioning (except for Grade 3 nausea, vomiting, diarrhea, or constipation).
* No significant change in clinical status that would, in the opinion of the investigator, increase the risk of adverse events associated with CIML NK infusion, (e.g., significant hypoxemia, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia)
* No evidence of active, uncontrolled infection. Patients receiving antibiotics for an infection may be treated if they have clinically responded to antibiotics. These cases should be reviewed with the study PI before proceeding.
* No systemic steroid therapy (oral or IV) of > 10mg prednisone or equivalent dose of other steroid agent on the day of NK cell infusion

If any of the above criteria are noted at these time points, please discuss with PI the benefits/risks of proceeding with the CIML infusion and document rationale for course of action taken in study regulatory binder. However, patient may still receive CIML NK infusion if relevant parameters are reviewed and both PI and IND holder agree with proceeding.

If inclusion/exclusion criteria are not met on planned day of CIML NK cell infusion, the NK cell infusion may be delayed for up to 24 hours to enable inclusion criteria to be met.

Criteria to Receive Venetoclax

* Adequate organ function within 24 hours of venetoclax initiation as defined below:

  * Total bilirubin: ≤1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then < 3 x ULN)
  * AST(SGOT)/ALT(SGPT): ≤3 x institutional ULN
  * No Grade ≥3 non-hematologic toxicities of cyclophosphamide and fludarabine conditioning (except for Grade 3 nausea, vomiting, diarrhea, or constipation).
* No significant change in clinical status that would, in the opinion of the investigator, increase the risk of adverse events associated with venetoclax administration, (e.g., significant hypoxemia, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, severe ongoing tumor lysis syndrome)
* No evidence of active, uncontrolled infection. Patients receiving antibiotics for an infection may be treated if they have clinically responded to antibiotics. These cases should be reviewed with the study PI before proceeding.
* No live vaccines within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Observing window is from Day 0 (day of CIML NK cell infusion) to Day +28
  A DLT is defined as an adverse event (AE) that is related to the CIML NK cell infusion with venetoclax as consolidation therapy. Toxicities are to be assessed according to the CTCAEv5.
Maximum Tolerated Dose (MTD) | Observing window is from Day 0 (day of CIML NK cell infusion) to Day +28
  The MTD in the CIML NK cell infusion with venetoclax as consolidation therapy is determined by the number of participants who experience a DLT. See previous primary outcome measure for the DLT definition. If ≤1 DLTs are observed at dose-level 0, this dose will be the MTD. If ≥2 DLTs are observed in a cohort of 5 evaluable participants, then the MTD is considered exceeded. If this is dose level 0, dose de-escalation will take place, and 5 evaluable participants will be enrolled at dose level -1. If ≥2 DLTs are observed at dose level -1, accrual will stop.

SECONDARY OUTCOMES:
Measurable Residual Disease Negative (MRD-) Rate | At +28 days post CIML NK Infusion
  MRD- rate is defined as the proportion pf participants achieving MRD. MRD clearance is evaluated by both highly sensitive flow cytometry and duplex sequencing on paired bone marrow samples.
100-day Leukemia-Free Survival (LFS) | 100 Days
  Leukemia free survival based on the Kaplan-Meier method is defined as the the duration of time from study entry to documented disease progression (leukemic relapse or death from any cause) or death. 100-day LFS is calculated from the KM curve with standard error.
1-year Leukemia-Free Survival (LFS) | 1 Year
  Leukemia free survival based on the Kaplan-Meier method is defined as the the duration of time from study entry to documented disease progression (leukemic relapse or death from any cause) or death. 1-year LFS is calculated from the KM curve with standard error.
100-day Overall Survival (OS) | 100 Days
  100-day OS is a probability estimated using the Kaplan-Meier method; OS is defined as the time from study entry to death, or censored at date last known alive.
1-year Overall Survival (OS) | 1 Year
  1-year OS is a probability estimated using the Kaplan-Meier method; OS is defined as the time from study entry to death, or censored at date last known alive.
Acute GVHD Rate | 1 Year
  Acute GVHD Rate is defined as the proportion of participants that has achieved acute GVHD. The criteria of acute GVHD grading is attached in protocol appendix c.
1-year Chronic GVHD Rate | 1 Year
  Chronic GVHD Rate is defined as the proportion of participants that has achieved chronic GVHD by NCI common toxicity criteria (appendix d).

CONTACTS AND LOCATIONS:
Overall Officials: Evan Chen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu